CLINICAL TRIAL: NCT00672516
Title: Management of Excessive Bleeding Following Cardiopulmonary Bypass: A Pilot Feasibility Study
Brief Title: Management of Bleeding Following Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Johns Hopkins University (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: 0604M85353; 20100962-A1
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hemorrhage; Cardiopulmonary Bypass
Keywords: hemorrhage; cardiopulmonary bypass; blood component transfusion; hemostasis, surgical
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We believe ongoing bleeding during complex cardiac surgery can be accurately measured and that administration of a specific blood product replacement strategy designed to optimally slow or stop the bleeding can be followed by the during the operation.

Patients at risk of significant bleeding after complex cardiac surgery will be approached to allow their operation to be watched by study personnel to see if ongoing blood loss can be accurately measured and to see how quickly a prescribed, standardized blood product replacement protocol to control the bleeding does slow or stop the bleeding. Permission to review the medical record to see if bleeding risk features can be identified and permission to follow the patient after surgery to see how they recover is also requested.

ELIGIBILITY:
Inclusion Criteria:

Eligible male and female patients will include those who are over 18 kg (identified as the lower inclusion threshold so as to standardize CPB circuit dilution) and less than 75 years old (to limit excessive stroke risk) and at theoretically increased risk for excessive bleeding following cardiopulmonary bypass, including patients:

1. undergoing repeat sternotomy, or
2. undergoing combined procedures (i.e. - valve and coronary artery surgery), or
3. undergoing multiple valve surgery, or
4. undergoing aortic root replacement with/without deep hypothermic circulatory arrest, or
5. undergoing complex congenital cardiac surgery

Exclusion Criteria:

Ineligible patients include those:

1. with known coagulation factor deficiency, or
2. refusing to receive donor blood products if necessary, or
3. undergoing emergency surgery, or
4. undergoing their first coronary artery bypass surgery or their first valve repair/replacement, or
5. with history of previous stroke or other significant thromboembolic event within 6 months (such as pulmonary embolism, valve obstruction [if not replacing this valve in upcoming operation], renal vein thrombosis, acute MI, DVT ), or
6. with known thrombophilia, or
7. with active infection (bacteremia, sepsis, endocarditis, meningitis, urinary tract infection, cholecystitis, cellulitis, pneumonia)
8. pregnant, or
9. weight > 150 kg or < 18 kg

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study populations includes male and female patients over 18 kg in weight and less than 75 years old who are undergoing cardiopulmonary bypass and are theoretically at risk for significant bleeding in the peri-operative period
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Tabulate the number of high risk subjects that must be screened and consented in order to find twenty subjects that meet the criteria of excessive bleeding following conventional therapy | end of trial
Determine blood loss, bleeding rate and blood transfusion prior to and following completion of algorithm-guided conventional transfusion therapy,including measured loss, rate of loss, volume of transfusion | During and immediately following completion of bypass OR in the first 24 hours after admission to the IUC, if significant bleeding occurs
Assess the relative accuracy and clinical relevance of measuring bleeding rate, blood loss and blood transfusion in the first 24 hours following designation of "excessive bleeding", including measured hourly outputs, rate of output and volume transfused | First 24 hours after operation
Assess the level of compliance to the Bleeding Management Algorithm | Immediate peri-operative period

SECONDARY OUTCOMES:
Tabulating adverse outcomes, including: 1) rate of re-exploration within the next 24 hours, 2) use of rescue therapeutics in accordance with local practice, and 3) mortality within 30 days | First 30 days post-operatively or until discharge, whichever comes first
Recording serious adverse events, such as myocardial infarction, thrombo-embolic events, etc. | First 30 days post-operatively or discharge, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Marie E Steiner, MD, MS, Study Chair — University of Minnesota; Philip Greilich, MD, Principal Investigator — University of Texas Souwthwestern Medical Center; Nauder Faraday, MD, Principal Investigator — Johns Hopkins Medical Center; Nigel S Key, MB, FRCP, Principal Investigator — University of North Carolina, Chapel Hill; Jerrold Levy, MD, Principal Investigator — Emory University
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Steiner ME, Despotis GJ. Transfusion algorithms and how they apply to blood conservation: the high-risk cardiac surgical patient. Hematol Oncol Clin North Am. 2007 Feb;21(1):177-84. doi: 10.1016/j.hoc.2006.11.009. PMID 17258126
- [Background] Levy JH, Tanaka KA, Steiner ME. Evaluation and management of bleeding during cardiac surgery. Curr Hematol Rep. 2005 Sep;4(5):368-72. PMID 16131437
- [Background] Avidan MS, Alcock EL, Da Fonseca J, Ponte J, Desai JB, Despotis GJ, Hunt BJ. Comparison of structured use of routine laboratory tests or near-patient assessment with clinical judgement in the management of bleeding after cardiac surgery. Br J Anaesth. 2004 Feb;92(2):178-86. doi: 10.1093/bja/aeh037. PMID 14722166